CLINICAL TRIAL: NCT01431651
Title: Asian Pacific Weight Loss and Metabolic Surgery Center
Brief Title: Probiotics Improve Gastrointestinal Symptoms After Roux-en-Y Gastric Bypass: A Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Principal Investigator, WEI-CHENG YAO, Min-Sheng general hospital IRB, Min-Sheng General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MSIRB2011010
Record Dates: First submitted 2011-09-01; First posted 2011-09-09 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Morbid Obesity
Keywords: Food and beverages; Food; Dietary supplements
MeSH Terms: conditions — Obesity, Morbid | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- probiotic, lifestyle counseling (Experimental)
  Interventions: Dietary Supplement: probiotics,digestive enzyme

INTERVENTIONS:
Dietary Supplement: probiotics,digestive enzyme — patients was randomized into 3 groups: clostridium butyricum MIYAIRI group (80 mg daily) bifidobacterium Longum BB536 group (2 packs daily) biotase:4 tables per day

SUMMARY:
Obesity has been a global epidemic. Currently, bariatric surgery has been recognized as the only successful treatment for morbid obesity. Laparoscopic gastric bypass (LGB) is the leading bariatric surgery worldwide including Taiwan, it's resulted in significant weight loss and resolution of metabolic co-morbidities in morbidly obese patients .

However, annoyed Gastro-Intestinal (GI) symptoms are a common complaint after gastric bypass like foul smell flatus, oil flatus and over flatus. The aim of this study was to determine whether probiotics would improve annoyed GI symptoms after gastric bypass.

Probiotics are live microorganisms (in most cases, bacteria) that are similar to beneficial microorganisms found in the human gut. They are also called "friendly bacteria" or "good bacteria." Probiotics are available to consumers mainly in the form of dietary supplements and foods.

DETAILED DESCRIPTION:
Probiotics are available in foods and dietary supplements (for example, capsules, tablets, and powders) and in some other forms as well. Examples of foods containing probiotics are yogurt, fermented and unfermented milk, miso, and some juices and soy beverages. In probiotic foods and supplements, the bacteria may have been present originally or added during preparation. In this study, we investigate the efficacy of probiotics for alleviating the annoyed GI symptoms after LGB.

Clostridium butyricum Probiotics is a novel microecological feed additive, it has the characteristic of heat tolerance, acid tolerance and antibiotic resistance and is general used to treat the intestinal tract disease in the clinical treatment. Its potential function in the situation that feed has been added universally with antibiotics will make it have a good development.

This randomized, placebo-controlled, double blind, prospective clinical trial was conducted among 60 patients undergoing gastric bypass for morbid obesity who had annoyed GI symptoms. Patients were randomized to the clostridium butyricum MIYAIRI group (80 mg daily , n=20,), bifidobacterium Longum BB536 group (2 packs daily, n=20),and biotase group(4 tablets daily, n=20). Control group (Biotase per day). Quality of life was measured and compared by the gastro-intestinal quality of life index (GIQLI) before and two weeks after in both groups. The higher score means that they have better quality of life. Through this study, we hope that we can find a effective probiotics can help all the patient received gastric bypass and bothered by their gastrointestinal problems also can improve their satisfaction of this operation.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity patients after gastric bypass with annoyed intestinal symptoms

Exclusion Criteria:

* cannot obey the orders to take medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Questionnaire of gastrointestinal quality of life | two weeks after taken drugs

CONTACTS AND LOCATIONS:
Overall Officials: YAO W C, Phd, Study Director — MSIRB
Locations (1):
- WJ Lee, Taoyuan, Taoyuan County, Taiwan